CLINICAL TRIAL: NCT04985123
Title: A Study on the Safety and Effectiveness of Subcutaneous Silicone Penile Implant Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: International Medical Devices, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00036006
Record Dates: First submitted 2021-07-16; First posted 2021-08-02 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Penile Implant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Silicone Block patients: All subjects who received a successful penile implantation with the Silicone Block by the surgeons at the centers in this study.
  Interventions: Device: Pre-Formed Penile Silicone Block Implant

INTERVENTIONS:
Device: Pre-Formed Penile Silicone Block Implant — Implantation of Pre-Formed Penile Silicone Block Implant

SUMMARY:
This study will identify a patient population who wishes to address a variety of concerns about the size, shape, or appearance of their penis with the placement of a subcutaneous Silicone Block Penile Implant. Because the Silicone Block is placed subcutaneously, the device can provide immediate and permanent improvements to the appearance of a man's penis. The most notable improvements are enhanced penile cosmesis, improved penile girth, and improved exposure of the penile shaft outside the plane of the body.

The plan is to conduct a study to examine the outcomes of this procedure with respect to:

* Incidences of adverse events
* Changes in flaccid penile length (through physical measurements pre and post-operatively in a consistent manner)
* Changes in flaccid penile girth (through physical measurements pre and post-operatively in a consistent manner)
* Changes in satisfaction scores with respect to penile size and patient self-confidence/self-esteem (through validated questionnaires)

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include men who are over 18 and under 65, circumcised, who have the perception of inadequate penile girth or appearance of length of penis, or penile deviation from straight plane in flaccid condition for whatever reason. Etiologies may include:
* A retractile penis or "buried penis" from infrapubic pannus
* A loss of length following radical prostatectomy or other trauma
* Congenital or acquired (e.g., Peyronie's Disease) mild curvature of the penis with indentation deformity and with curvature less than 30 degrees with no plan to have other corrective procedures (e.g. surgery, intralesional injection of collagenase clostridium histolyticum)
* Patient perception of a penis of inadequate size and patient desire for cosmetic enhancement

Exclusion Criteria:

* Men who are unable to give informed consent
* An uncircumcised penis
* Micro-penis (stretched flaccid penile length <6cm)
* Prior penile girth enhancement procedure of any sort, including grafts or subcutaneous injections, previous Xiaflex injection
* History of immunosuppression and/or HIV
* Men who are on anti-coagulation medication which cannot be stopped
* Uncontrolled diabetes
* Active genitourinary skin infection
* History of recurrent or active urinary tract infection (UTI)
* Patients unwilling to comply with post-operative instructions
* Patients who smoke and are unwilling to stop 2 weeks before surgery and for at least 6 weeks after surgery.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects who received a successful penile implantation with the Silicone Block by the surgeons at the centers in this study.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-07-30 (Actual); Primary Completion 2023-05-25 (Estimated); Study Completion 2023-05-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events as Assessed by Observation | 8 weeks
Incidence of Adverse Events as Assessed by Observation | 3 months

SECONDARY OUTCOMES:
Size of Flaccid Penile Girth as Measured by Physicians | 8 weeks
Size of Flaccid Penile Girth as Measured by Physicians | 3 months
Patient Reported Satisfaction as Assessed by Validated Questionnaires | 8 weeks
Patient Reported Satisfaction as Assessed by Validated Questionnaires | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Uropartners, Chicago, Illinois, United States